CLINICAL TRIAL: NCT00002228
Title: A Phase II Evaluation of the Safety, Plasma Pharmacokinetics, and Antiviral Activity of T-20 Administered to HIV-1 Positive Adults By Continuous Subcutaneous Infusion or Subcutaneous Injection
Brief Title: A Study of T-20 in HIV-Positive Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Trimeris (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 295A; TRI-003
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1999-04

CONDITIONS: HIV Infections
Keywords: Injections, Subcutaneous; HIV-1; Anti-HIV Agents; peptide T20
MeSH Terms: conditions — HIV Infections | interventions — Enfuvirtide

INTERVENTIONS:
Drug: Enfuvirtide

SUMMARY:
The purpose of this study is to see if it is safe and effective to give T-20 to HIV-positive adults. T-20 is an anti-HIV drug.

DETAILED DESCRIPTION:
Patients are randomly placed into 1 of 6 groups: 4 dose levels of T-20 are given by subcutaneous infusion and 2 by subcutaneous injection. The entire study lasts 7 weeks; including a 2-week screening period, followed by 28 days of treatment and 1 week of follow-up.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Any antiretroviral agent, provided the regimen has not changed within 6 weeks of the screening visit.
* Antibiotics for bacterial infections.
* Prophylactic medications for P. carinii pneumonia and for M. avium, including azithromycin.
* Medications for symptomatic treatment such as antipyretics, analgesics, and antiemetics.

Patients must have:

HIV-1 seropositive status.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

Concurrent neoplasm (except for basal cell carcinoma of the skin, in situ carcinoma of the cervix, and non-disseminated stable Kaposi's sarcoma).

Concurrent Medication:

Excluded:

* Patients must not be taking any concurrent antiretroviral therapy (for at least 2 weeks prior to baseline) or the patient is to be on a stable antiretroviral regimen which has not changed for at least 6 weeks prior to baseline.
* Treatment with any of the following:
* immunomodulators, biological response modifiers, chemotherapy that cannot be discontinued for the duration of the study, astemizole, terfenadine, cisapride, triazolam, midazolam, rifampin, clarithromycin, or an investigational drug within 30 days prior to the initial visit.

Patients with the following prior conditions are excluded:

* Evidence of active opportunistic infections, or unexplained temperature greater than or equal to 38.5 Celsius for 7 consecutive days within 30 days prior to screening visit.
* Chronic diarrhea (defined as greater than 3 liquid stools per day which persists for 15 days) within 30 days prior to screening visit.
* Diagnosis of hemophilia or other clotting disorders.

Prior Medication:

Excluded:

- Prior treatment with an HIV vaccine.

Prior Treatment:

Excluded:

Major organ allograft.

Risk Behavior:

Excluded:

Evidence of substance abuse or addiction that, in the opinion of the investigator, may interfere with the patient's ability to comply with the dosing schedule and protocol evaluations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78

CONTACTS AND LOCATIONS:
Overall Officials: Sam Hopkins, Study Chair
Locations (11):
- United States (11):
  - Univ of Alabama at Birmingham / 1917 AIDS O/P Cln, Birmingham, Alabama
  - UCLA School of Medicine / Ctr for Research and Education, Los Angeles, California
  - San Francisco Gen Hosp, San Francisco, California
  - Quest Clinical Research, San Francisco, California
  - IDC Research Initiative, Altamonte Springs, Florida
  - Northwestern Univ / Infect Dis Div / Pasavant Pav 828, Chicago, Illinois
  - Johns Hopkins Hosp, Baltimore, Maryland
  - CRI of New England, Brookline, Massachusetts
  - NYU Med Ctr / C & D Building, New York, New York
  - Univ North Carolina at Chapel Hill / Dept of Medicine, Chapel Hill, North Carolina
  - Univ of Texas / Thomas Street Clinic, Houston, Texas